CLINICAL TRIAL: NCT01112319
Title: The Effects of the Electro, Heat and Cold -Therapy During Physiotherapy Treatment in OA of KNEE - Prospective Randomize Trial
Brief Title: The Effects of the Electro, Heat and Cold -Therapy During Physiotherapy Treatment in Osteoarthritis(OA) of KNEE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: not patient recruitment
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 041-2010
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Knee Pain; Osteoarthritis
Keywords: COLD HOT or Electrotherapy treatment
MeSH Terms: conditions — Osteoarthritis | interventions — Control Groups

ARMS (2):
- Elf_care (Experimental): The trial group will receive with Elf_Care unit (Hot-Cold & Electrotherapy) during physiotherapy treatment ( 28 minutes twice a week)
  Interventions: Device: Elf care
- control group (Active Comparator): The control group will receive before physiotherapy COLD HOT or Electrotherapy treatment depends on the patient and physiotherapy prefer.
  Interventions: Other: control group

INTERVENTIONS:
Device: Elf care — elfcare device
  Arms: Elf_care
Other: control group — regular physiotherapy treatment
  Arms: control group

SUMMARY:
The objective of this clinical trial is to evaluate the pain relief and daily functioning improve, in patients suffering of Osteoarthritis of knee, with HOT/COLD/ Electro therapy during physiotherapy treatment

DETAILED DESCRIPTION:
Prospective randomize trial. The patients with knee pain and osteoarthritis, that were referred to the physiotherapy treatment.

Each patient will be checked twice by the physiotherapy team, in the first and in the last physiotherapy treatment. Test muscle strength of QUADRICEPS, GLUTEOUS MEDIUS and HAMSTRING will be measured by Dynamometer (the dynamometer expressed in a quantitative way the muscle force) The population will randomized separated in trail and control group. The control group will receive before physiotherapy COLD HOT or Electrotherapy treatment depends on the patient and physiotherapy prefer.

The trial group will receive with Elf_Care unit (Hot-Cold & Electrotherapy) during physiotherapy treatment ( 28 minutes twice a week) The protocol treatment includes 28 minutes of cycling cold/hot/cold/hot treatment (2*7 min cold: 10…15 degrees; 2*7 min hot: 39..42 degrees,). During this 28 minutes the patient also receive tolerable intensity Premodulated Interferential current with sweep Beat frequency (3Hz…200Hz), Carrier frequency 5kHz ; Electrodes setup: Thermo Electrode and 2 Regular Electrodes After the treatment the control and trail group will evaluate with 0-10 visual analogue scale VAS, Oxford Knee Score and WOMAC The population will receive treatment twice a week for one month.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients more than 60 years old
* Patients suffering from knee pain due to osteoarthritic changes in radiographic plains.
* Patients in medical condition to receive physiotherapy treatment
* Patients who are willing to participate in the trial, to come to all scheduled visits and to sign the informed consent forms.

Exclusion Criteria:

* Patients receiving other methods of treatment to this area,
* Patients with concomitant other injury of the knee.
* Dermatological affection with contraindication use of hot, cold and/or electrical stimulation
* Non cooperative patient with the basic rehab program.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
The effects of the electro, heat and cold -therapy during physiotherapy treatment | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel